CLINICAL TRIAL: NCT01043640
Title: Allogeneic Hematopoietic Stem Cell Transplantation for Standard Risk Inherited Metabolic Disorders
Brief Title: Allogeneic Bone Marrow Transplant for Inherited Metabolic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS088; MT2009-19 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-09

CONDITIONS: Mucopolysaccharidosis; Hurler Syndrome; Hunter Syndrome; Maroteaux-Lamy Syndrome; Sly Syndrome; Alpha Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Adrenoleukodystrophy (ALD); Krabbe Disease; Metachromatic Leukodystrophy (MLD); Sphingolipidoses; Peroxisomal Disorders
Keywords: inherited metabolic disorders
MeSH Terms: conditions — Mucopolysaccharidoses; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; alpha-Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Adrenoleukodystrophy; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Sphingolipidoses; Peroxisomal Disorders | interventions — Alemtuzumab; Cyclophosphamide; Busulfan; Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Patients (Experimental): Includes patients who received allogeneic stem cell transplantation following treatment plan of Campath-1H, cyclophosphamide, cyclosporine A, mycophenolate mofetil, and busulfan.
  Interventions: Drug: Campath-1H; Drug: Cyclophosphamide; Drug: Busulfan; Procedure: Allogeneic stem cell transplantation; Drug: Cyclosporine A; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Campath-1H — Administered Days -21, -20 and -19, 0.3 mg/kg subcutaneously (SQ) or intravenously (IV)
  Other Names: Alemtuzumab
Drug: Cyclophosphamide — Administered days -10 through -6, 50 mg/kg/day intravenous (IV) over 2 hours - with Mesna continuous infusion or 5 times daily.
  Other Names: Cytoxan(R)
Drug: Busulfan — Administered every 6 hours: If < or = 12 kg then 1.1 mg/kg/dose intravenous (IV). If > 12 kg then 0.8 mg/kg/dose IV
  Other Names: Busulfex(R)
Procedure: Allogeneic stem cell transplantation — Administered > 24 hours after last dose of busulfan.
  Other Names: stem cell transplant
Drug: Cyclosporine A — 2.5 mg/kg/dose intravenous (IV_ beginning on day -3. Frequency of daily dosing will be based on the recipient's body weight:
  * If body weight is ≤ 40 kg dosing will be 3 times daily
  * If body weight is > 40 kg dosing will be 2 times daily An attempt will be made to maintain a trough cyclosporine level of 250 mg/L to 350 mg/L. Once the patient can tolerate oral medications and has a normal gastrointestinal transit time, CsA will be converted to an oral form at a dose 2 times the current IV dose (maximum 12.5 mg/kg/day as initial oral dose).
  Other Names: CsA
Drug: Mycophenolate Mofetil — 15 mg/kg/dose (max dose of 1gram) IV three times a day beginning on Day -3 at a dose based on body weight: The same dosage is used orally or intravenously. Stop MMF at day +42 or 7 days after engraftment achieved (ANC>500 x 10^6 neutrophils/L x 3 days and chimerism >90%), whichever is later.
  Other Names: MMF

SUMMARY:
Rationale: Chemotherapy administration before a donor stem cell transplant is necessary to stop the patient's immune system from rejecting the donor's stem cells. When healthy stem cells from a donor are infused into the patient, the donor white blood cells can provide the missing enzyme that causes the metabolic disease. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving a monoclonal antibody, alemtuzumab, before transplant and cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening. This may be an effective treatment for inherited metabolic disorders.

Purpose: The design of this study is to achieve donor cell engraftment in patients with standard-risk inherited metabolic diseases with limited peri-transplant morbidity and mortality. This will be achieved through the administration of the chemotherapy regimen described. The intention is to follow transplanted patient for years after transplant monitoring them for complications of their disease and assisting families with a multifaceted interdisciplinary approach.

DETAILED DESCRIPTION:
Primary Objective:

* To estimate the proportion of patients with donor derived engraftment at day 100 post transplant as defined by 80% or greater donor cells in the CD3 (T cell) fraction

Secondary Objectives:

* To determine the incidence and severity of graft-versus-host disease (GVHD) by day 100
* To determine the incidence of peri-transplant mortality (death by day 100)
* To monitor donor cell chimerism at various time points following allogeneic transplantation with this transplant regimen as determined at day 28, 42, 100, 6 months and yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosis of one of the following: mucopolysaccharidosis disorder, glycoprotein metabolic disorder, sphingolipidoses or inherited leukodystrophy, peroxisomal disorder or other inherited diseases of metabolism
* Must have an acceptable graft source as defined by University of Minnesota criteria
* Adequate organ function

Exclusion Criteria:

* Pregnant - menstruating females must have a negative serum pregnancy test within 14 days of treatment start
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2009-12; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant Patients: Includes patients who received allogeneic stem cell transplantation following treatment plan of Campath-1H, cyclophosphamide, cyclosporine A, mycophenolate mofetil, and busulfan.
  Campath-1H: Days -21, -20 and -19, 0.3 mg/kg SQ or IV Cyclophosphamide: Days -10 through -6, 50 mg/kg/day IV with Mesna Busulfan: Days -5 through Day -2, 1.1 mg/kg/dose IV if ≤ 12 kg; 0.8 mg/kg/dose IV if > 12 kg Allogeneic stem cell transplantation: > 24 hours after last dose of busulfan Cyclosporine A: 2.5 mg/kg/dose IV beginning on day -3. Dosing will be 3 times daily if body weight is ≤ 40 kg and 2 times daily if body weight is > 40 kg
  Mycophenolate Mofetil: 15 mg/kg/dose (max dose of 1gram) IV three times a day beginning on Day -3 at a dose based on body weight:
  Stop MMF at Day +42 or 7 days after engraftment achieved (ANC>500 x 10^6 neutrophils/L x 3 days and chimerism >90%), whichever is later.
Period: Overall Study
Arm/Group | Transplant Patients
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Donor Derived Engraftment
Description: Donor derived engraftment is defined as 80 percent or greater donor cells in the recipient's bone marrow and blood cells.
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 42

2. Secondary Outcome: Number of Patients With Grade 0 Graft-Versus-Host Disease (GVHD)
Description: GVHD grading is performed using modified Glucksberg criteria and is as follows:
  grade 0: absence of any skin, liver and/or gastrointestinal (GI) involvement grade 1: skin stage 1 or 2 only grade 2: skin stage 3 or liver stage 1 or lower GI stage 1 or upper GI involvement grade 3: skin stage 0 - 3 plus liver stage 2-4 or lower GI stage 2-3 grade 4: skin stage 4 or lower GI stage 4
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 32

3. Secondary Outcome: Number of Patients With Grade 1 Graft-Versus-Host Disease (GVHD)
Description: as for outcome 2
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 2

4. Secondary Outcome: Number of Patients With Grade 2 Graft-Versus-Host Disease (GVHD)
Description: as for outcome 2
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 5

5. Secondary Outcome: Number of Patients With Grade 3 Graft-Versus-Host Disease (GVHD)
Description: as for outcome 2
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 2

6. Secondary Outcome: Number of Patients With Grade 4 Graft-Versus-Host Disease (GVHD)
Description: as for outcome 2
Time Frame: Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 5

7. Secondary Outcome: Number of Patients Who Died Peri-Transplant
Description: Peri-transplant is defined as within 100 days of transplant.
Time Frame: By Day 100 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
Participants | 2

8. Secondary Outcome: Donor Cell Chimerism Following Transplant
Description: Donor cell chimerism is defined as the percentage of bone marrow and blood cells in the recipient that are of donor origin.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
percentage of donor cells | 95 (9)

9. Secondary Outcome: Donor Cell Chimerism Following Transplant
Description: as for outcome 8
Time Frame: Day 42
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
percentage of donor cells | 93 (15)

10. Secondary Outcome: Donor Cell Chimerism Following Transplant
Description: as for outcome 8
Time Frame: Day 100
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
percentage of donor cells | 90 (26)

11. Secondary Outcome: Donor Cell Chimerism Following Transplant
Description: as for outcome 8
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
percentage of donor cells | 94 (22)

12. Secondary Outcome: Donor Cell Chimerism Following Transplant
Description: as for outcome 8
Time Frame: One year
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Transplant Patients
Number analyzed (Participants) | 46
percentage of donor cells | 99 (4)

ADVERSE EVENTS:
Arm/Group | Transplant Patients
Serious Adverse Events (participants affected / at risk) | 8/46
Other Adverse Events (participants affected / at risk) | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant Patients (N=46)
Pericardial Effusion (Cardiac disorders) | 2
Renal Failure (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Veno-Occlusive Disease (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Intracerebral Hemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant Patients (N=46)
Anorexia (Metabolism and nutrition disorders) | 7
Bilirubin Increased (Investigations) | 16
Diarrhea (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Fever (General disorders) | 11
Graft Versus Host Disease (General disorders) | 9
Headache (Nervous system disorders) | 3
Hemorrhage, Gastrointestinal (Gastrointestinal disorders) | 8
Hemorrhage, Genitourinary (Renal and urinary disorders) | 10
Hives (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 21
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14
Infection, NOS (Infections and infestations) | 35
Infection, Respiratory (Infections and infestations) | 9
Mucositis (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 6
Pericardial Effusion (Cardiac disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 10
Tachycardia (Cardiac disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Infection, Gastrointestinal (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No